CLINICAL TRIAL: NCT01181037
Title: Bipolar H.A Versus Trochanteric Antegrade Nail for Treatment of Displaced Subcapital Femoral Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: mmc10039-2010ctil; 0392010
Record Dates: First submitted 2010-05-02; First posted 2010-08-13 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Displaced Subcapital Femoral Fracture
Keywords: Displaced subcapital femoral fracture; Bbipolar H.A.; CRIF with Ttrochanteric Antegrade Nail

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 100 patients, displaced subcapital fracture, T.A.N nail.: 100 patients sustained a displaced femoral subcapital fracture, that were operated on with closed reduction and internal fixation with TAN nail.
- 100 patients, displaced subcapital fracture, Bipolar H.A..

SUMMARY:
A retrospective study to compare clinical results of patients that were treated by Bipolar H.A. vs. closed reduction and internal fixation with Trochanteric Antegrade Nail for displaced femoral subcapital fracture.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral subcapital fracture.
* Active patient.
* Age 40-85.
* Patient was treated by one of the two methods.

Exclusion Criteria:

* Age out of range.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients sustained a displaced subcapital femoral fracture and were operated on by colsed reduction and internal fixation with T.A.N nail or Bipolar hemiarthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
describe treatment of patients that were treated by Bipolar H.A. vs. closed reduction and internal fixation | 6month to 3 years following operation
  A retrospective study will defer between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel